CLINICAL TRIAL: NCT04499703
Title: Evaluation of the Retinal Health Monitoring System - Retinal Thickness Module in Subjects With Normal Macular Thickness and Subjects With Center-involving Macular Edema
Brief Title: Evaluation of the Retinal Health Monitoring System Thickness Module
Status: Completed | Type: Observational
Sponsor: Kubota Vision Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SCT-202 D
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Macular Edema; Macular Degeneration
Keywords: Age-Related Macular Degeneration; macular edema; retinal vein occlusion; diabetic macular edema
MeSH Terms: conditions — Macular Edema; Macular Degeneration; Retinal Vein Occlusion | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: Subjects with normal macular thickness in one or both eyes.
  Interventions: Device: RHMS-RTM; Diagnostic Test: SD-OCT
- Group 2: Subjects with center-involving macular edema due to wAMD in one or both eyes
  Interventions: Device: RHMS-RTM; Diagnostic Test: SD-OCT
- Group 3: Subjects with center-involving macular edema due to DR or RVO in one or both eyes
  Interventions: Device: RHMS-RTM; Diagnostic Test: SD-OCT

INTERVENTIONS:
Device: RHMS-RTM — Assessment of retinal thickness
  Other Names: Handheld swept source (SS) optical coherence tomography (OCT)
Diagnostic Test: SD-OCT — Assessment of retinal structure

SUMMARY:
Evaluate the ability and accuracy of the Retinal Health Monitoring System - Retinal Thickness Module (RHMS - RTM).

DETAILED DESCRIPTION:
Evaluation of the Retinal Health Monitoring System - Retinal Thickness Module in subjects with normal macular thickness and subjects with center-involving macular edema.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥50.
2. Corrected visual acuity (VA) of 20/125 or better, in the study eye(s)
3. Media clarity, undilated pupil size, and subject cooperation sufficient to obtain adequate OCT B-scans in the study eye(s)
4. Able to perform self-testing of retinal thickness with the RHMS-RTM after training
5. Able and willing to provide written informed consent before undergoing any study-related procedures
6. Group 1: Macula with normal thickness [central subfield thickness (CST): <305μm in women, and <320μm in men as measured by Heidelberg Spectralis SD-OCT in at least one eye. Patients diagnosed with dry AMD are eligible for enrollment into Group 1. No history of wAMD, DR, or RVO in either eye
7. Group 2 and Group 3, in at least one and the same eye: History of center-involving macular edema due to wAMD (Group 2); or DR or RVO (Group 3); Macular edema on SD-OCT with CST ≥305 μm in women, and ≥320μm in men as measured by Heidelberg Spectralis SD-OCT.

Exclusion Criteria:

1. History of corneal refractive surgery [e.g., laser-assisted in situ keratomileusis (LASIK), photorefractive keratectomy (PRK), radial keratotomy (RK)] in the study eye(s)
2. History of epiretinal membrane, vitreomacular traction, or macular hole in the study eye(s)
3. Participation in any study using an investigational drug within 30 days of screening or an investigational device within 60 days of screening
4. Refractive error within defined limits
5. History of photocoagulation laser scar or other retinal scar in the central 3 mm of the macula, in the study eye(s)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects aged ≥ 50 years old with normal macular thickness, center-involving macular edema due to wAMD, diabetic retinopathy or retinal vein occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2021-01-25 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Evaluation of the RHMS-RTM retinal thickness measurements | 1 day
  To evaluate the ability of the RHMS-RTM device to measure retinal thickness

SECONDARY OUTCOMES:
Repeatability of RHMS-RTM retina thickness measurements | 1 day
  To assess repeatability of the RHMS-RTM device
Comparison of retinal thickness measurements between the RHMS-RTM and the SD-OCT | 1 day
  To evaluate the agreement of measurements by the RHMS-RTM and SD-OCT
Intraretinal and subretinal fluid detection | 1 day
  To evaluate the feasibility of intra- and sub-retinal fluid detection

CONTACTS AND LOCATIONS:
Overall Officials: Marion Munk, MD, PhD, Principal Investigator — Inselspital, University Hospital Bern
Locations (1):
- Inselspital, University Hospital Bern, Department of Ophthalmology, Bern, Switzerland